CLINICAL TRIAL: NCT05838430
Title: The Effects of Solriamfetol and CBT-I (Alone and in Combination) on Sleep Continuity, Sleepiness, Fatigue, and Performance in Patients With Insomnia Disorder
Brief Title: Solriamfetol and CBT-I in Patients With Insomnia Disorder
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Axsome Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 850945
Record Dates: First submitted 2023-03-06; First posted 2023-05-01 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Insomnia
Keywords: Insomnia; Medication; Fatigue; Performance; CBT-I
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Fatigue | interventions — solriamfetol; Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: A 2x2 mixed model design. The two factors will be 1) treatment (+/- solriamfetol and +/- CBT-I) and 2) Time (pre-post assessment, with additional follow-up data).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding only applies to the medication arm. The randomization schedule was developed by our statistician and sent directly to research pharmacy for implementation.
  The four arms are as follows:
  1. Solriamfetol + CBT-I
  2. Placebo + CBT-I
  3. Solriamfetol Only
  4. Placebo Only
  All conditions engage in monitoring and assessment.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Solriamfetol+ CBT-I (Experimental)
  Interventions: Drug: Solriamfetol 75 MG; Behavioral: Cognitive Behavioral Therapy for Insomnia (CBT-I)
- Solriamfetol Only (Experimental)
  Interventions: Drug: Solriamfetol 75 MG; Other: Monitoring
- Placebo + CBT-I (Active Comparator)
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia (CBT-I); Other: Placebo
- Placebo Only (Placebo Comparator)
  Interventions: Other: Monitoring; Other: Placebo

INTERVENTIONS:
Drug: Solriamfetol 75 MG — Solriamfetol (trade name Sunosi), is a norepinephrine-dopamine reuptake inhibitor available in 75mg and 150mg tablets for oral administration during the day. Solriamfetol's primary indication is to treat excessive daytime sleepiness (EDS) in patients diagnosed with obstructive sleep apnea or Narcolepsy. It binds to the dopamine and the norepinephrine transporters with affinities (Ki) of 14.2 μM and 3.7 μM, respectively),does not undergo significant metabolism in humans, and has a Tmax of ~2 hours (range 1.25-3.0 hours) and a T1/2 of ~7.1 hours.
  Arms: Solriamfetol Only; Solriamfetol+ CBT-I
Behavioral: Cognitive Behavioral Therapy for Insomnia (CBT-I) — Treatment will be conducted via a HIPAA compliant video link (Zoom). Sessions 1-8 will follow our published protocol (published in 2005 by Springer).
  Each session will be conducted individually and have a singular focus per session.
  All sessions following the delivery of sleep restriction therapy & stimulus control instructions (post Session 2) will include, as needed, management of non-adherence and/or time-in-bed titration.
  Arms: Placebo + CBT-I; Solriamfetol+ CBT-I
Other: Monitoring — No CBT-I will be administered, however, the tracking system used for CBT-I will be used for all subject conditions. This includes a sleep disorder symptoms screener, the administration of several questionnaires on a weekly basis, and the administration of daily sleep diaries online or via iPhone. Note: it is a common effect that regular monitoring of this type produces perceived clinical benefit.
  Arms: Placebo Only; Solriamfetol Only
Other: Placebo — Placebo, identical in appearance to the active drug.
  Arms: Placebo + CBT-I; Placebo Only

SUMMARY:
Medication is FDA approved. The objective of this project is to test the efficacy of solriamfetol for treating insomnia (alone and in combination with Cognitive Behavioral Therapy for Insomnia [CBT-I]). Ultimately, this study will test whether wake extension (regardless of how it is achieved) will consolidate sleep and improve sleep continuity.

DETAILED DESCRIPTION:
The current proposal is for a one-year study to investigate whether solriamfetol can improve sleep continuity and daytime performance, alone and in combination with Cognitive Behavioral Therapy for Insomnia. It is expected (given a common mechanism [wake extension]) that both Cognitive Behavioral Therapy for Insomnia and treatment with solriamfetol will improve sleep continuity, and that such effects will potentially be additive.

ELIGIBILITY:
Inclusion Criteria:

• Participants will meet the diagnostic criteria for Insomnia Disorder according to Diagnostic and Statistical Manual of Mental Disorders (DSM-5).

In addition, the complaint of disturbed sleep will meet the following criteria:

* ≥ 30 minutes to fall asleep (SL) and/or ≥ 2 awakenings per night of ≥ 15 minutes duration and/or wake after sleep onset (WASO) time of ≥ 30 minutes where total sleep time (TST) did not exceed 6 hours (unless sleep efficiency [SE] is ≤ 80%).
* The problem is present for > 3 nights per week.
* The problem duration exceeds ≥ 6 months.
* The complaint of impaired daytime function must include, although not limited to, the report of daytime fatigue, sleepiness, or both.
* Preferred regular sleep phase between 10:00 PM and 8:00 AM
* Must garner physician's assent from their primary care clinician

Exclusion Criteria:

* Use of medication expressly for the purpose of falling or staying asleep (e.g., trazodone/ desyrel, melatonin, Tylenol PM, Nyquil, Benadryl).
* Night shift work
* Compromised renal function
* Major Coronary Artery Disease and/or uncontrolled (with meds) Hypertension
* Planning to become pregnant, pregnant, and/or breastfeeding
* Unstable medical or psychiatric illness
* Symptoms suggestive of sleep disorders other than insomnia
* Polysomnographic data indicating sleep disorders other than insomnia
* Evidence of active illicit substance use, abuse, or dependence
* Use of CNS active medications that are for treatment of insomnia or are thought to have caused insomnia as a side effect
* Inadequate language comprehension
* Current or past experience with CBT-I
* No access to the computers, I-Pads, or the internet

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07-31 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Sleep Continuity | End of Treatment (12 Weeks)
  Reflected by total wake time [time spent awake in bed] as measured via a web based self-report Sleep Diary. This variable is calculated by summing the estimates for sleep latency (SL), sleep after wake onset (WASO), and early morning awakening (EMA).

SECONDARY OUTCOMES:
Insomnia Severity | End of Treatment (12 Weeks)
  As measured by the Insomnia Severity Index. Range of scores = 0 to 28, with a higher score indicating more severe insomnia.
Daytime Sleepiness | End of Treatment (12 Weeks)
  As measured by the Epworth Sleepiness Scale. Range of scores = 0 to 24, with a higher score indicating more severe daytime sleepiness.
Fatigue | End of Treatment (12 Weeks)
  As measured by Fatigue Severity Scale. Range of scores = 9 to 63, with a higher score indicating more severe fatigue.
Adherence to "sleep rescheduling" | Throughout treatment (over 8 weeks)
  Sleep rescheduling is a core component of Cognitive Behavioral Therapy for Insomnia, and adherence to it will be measured by the difference between prescribed time to bed and time out of bed and actual time to bed and time out of bed as reported on daily sleep diary entries.
Daytime Function | End of Treatment (12 Weeks)
  As measured by Functional Outcomes of Sleep Questionnaire (FOSQ-10) Range of scores = 10-40, with lower scores indicating more severe daytime function impairment.
Mood Disturbance | End of Treatment (12 Weeks)
  Total Mood Disturbance Score on Profile of Mood States Range of scores = 0-20, with higher scores indicating more severe mood disturbance.
Alertness | Throughout treatment (over 8 weeks)
  As measured by average response time (milliseconds) on a Psychomotor Vigilance Test.
  Range of scores = 0 to 180000 milliseconds, with a higher score indicating lower levels of alertness.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Behavioral Sleep Medicine Program, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
The investigators do not plan on sharing IPD with other researchers.